CLINICAL TRIAL: NCT02564458
Title: Fitness in Allogeneic Stem Cell Transplantation
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William A. Wood, MD, Dr. William A. Wood, MD, MPH, UNC Lineberger Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1705; 1R21CA192127-01A1 (NIH)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interval Exercise Training/Motivational Accelerometry (IET/MA) (Experimental): All patients on the experimental arm receive the intervention of 5-12 weeks of pre-transplant IET, motivational accelerometry via the FitBit Surge, pre- and post-fitness assessments, and periodic quality of life and symptom surveys.
  Interventions: Behavioral: Interval Exercise Training/Motivational Accelerometry
- Normal Standard of Care (control) (No Intervention): All patients on the control arm participate in the pre- and post-fitness assessment, are given the FitBit Surge without the motivational component, and are also given periodic quality of life and symptom surveys.

INTERVENTIONS:
Behavioral: Interval Exercise Training/Motivational Accelerometry — During the 5-12 weeks before allogeneic stem cell transplant, the patient will participate in an at home, interval exercise training (IET) program, as well as wear a physical activity tracker, the FitBit Surge, combined with a weekly motivational call, termed Motivational Accelerometry (MA). The combined intervention is referred to as (IET/MA). The first week of the IET program consists of the participants being asked to engage in 30 minutes of aerobic exercise at any intensity for 3-4 days. For weeks two and beyond, patients be asked to undergo 3-4 sessions of IET, consisting of a 5 minute warm-up and five 2-minute intervals, with the goal of reaching 80% MHR, separated by 3 minutes of recovery/light activity in between each interval. Each exercise session is a total of 30 minutes. In addition, each week prior to transplant, the patient will receive a weekly check-in/motivational call from the study staff in order to track progress and motivate the patient to continue participation.
  Arms: Interval Exercise Training/Motivational Accelerometry (IET/MA)

SUMMARY:
Purpose: The primary hypothesis of this study is that the combination of interval exercise training (IET) as well as motivational accelerometry (MA) delivered both as a 5-12 week intervention that will improve cardiorespiratory fitness in patients preparing to undergo allogeneic hematopoietic cell transplantation (alloHCT). MA is not an established term, but in respect to this study, MA refers to the use of wearable accelerometry paired with regular intervals of physical activity coaching from members of the study staff during the IET training. The study will also look at several secondary endpoints including the association of the intervention with changes in cyclin-dependent kinase inhibitor 2A, multiple tumor suppressor 1 (p16INK4a), and the association of the intervention with changes in symptoms and quality of life before and after transplant.

Participants: 60 patients will be randomized into two groups, 30 in the intervention group consisting of both IET and MA, and 30 in the control group applying usual care and use of wearable accelerometry without motivational physical activity coaching.

Procedures (methods): Results of this study will inform a randomized, multi-site study of a pre-transplant exercise intervention.

DETAILED DESCRIPTION:
The investigator team for the current protocol has recently completed a single-arm pilot protocol (LCCC 1311) of a 6-week home-based unsupervised IET program (goal of three IET sessions per week, 65%-95% Max Heart Rate [MHR]) in patients planning to undergo alloHCT. In our study, participants preparing to undergo alloHCT experienced an average 3.8ml/kg*min improvement in peak volume of oxygen consumed (VO2peak) from pre to post-intervention. Patients in LCCC 1311 wore FitBit accelerometers throughout the study period.

The primary purpose of the current randomized controlled trial is to determine, in patients preparing to undergo alloHCT, whether an intervention comprised of interval exercise training and motivational accelerometry (IET/MA) will improve cardiorespiratory fitness more than the control group who receives usual care and an accelerometer without motivational physical activity coaching. The study will also look at several secondary endpoints including the association of the intervention with changes in p16INK4a, and the association of the intervention with changes in symptoms and quality of life before and after transplant.

This randomized controlled trial will include 60 patients preparing to undergo alloHCT (30 in the intervention group, 30 in the control group). We plan to analyze the effect of IET/MA on VO2peak. Subjects will be recruited after their transplant teams have determined that they will undergo alloHCT within the subsequent 5-12 weeks. Following recruitment, patients will undergo baseline fitness assessments consisting of cardiorespiratory exercise testing using indirect calorimetry on a cycle ergometry (for the assessment of VO2peak), 6 minute walk distance testing, and baseline physical activity, symptom and quality of life questionnaires. Participants randomized to the IET/MA group will then receive an individualized IET/MA prescription for a duration of at least 5 weeks, up until the time of admission for alloHCT or 12 weeks from the initiation of IET/MA, whichever occurs first. The mode of exercise can be walking, jogging, running, cycling, elliptical, stair climbing, or a combination of these, and will be performed unsupervised at home. For the first week, participants will be asked to engage in 30 minutes of aerobic exercise at any intensity for 3-4 days. For weeks two and beyond, participants will undergo 3-4 sessions of IET, consisting of a 5 minute warm-up and five 2-minute intervals, with the goal of reaching 80% MHR, separated by 3 minutes of recovery/light activity in between each interval. Each exercise session is a total of 30 minutes. Fitness assessments will be completed at the end of the intervention period, at the time of admission for alloHCT. Based on the improvement in VO2peak seen in the pre-alloHCT patient population in LCCC 1311, the current study is powered to detect a 3.8ml/kg*min VO2peak improvement in the intervention group relative to the control group.

All participants in both groups will be provided with a FitBit Surge accelerometer. Participants in the intervention group will also receive weekly motivation from a study team member to achieve a 10% week over week improvement in average steps/day. Participants in the control group will not receive this physical activity coaching. Participants will continue to wear the accelerometers after the intervention and until 1 year following alloHCT. Participants in both groups will have blood drawn for p16INK4a levels before and after the IET intervention. Participants in both groups will also complete symptom and quality of life questionnaires before the intervention and periodically throughout the year following alloHCT (please see study plan and time and events tables).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age, inclusive
* Verification of a functioning email address and access to electronic device(s) with the ability to charge and sync the FitBit Surge
* Planned allogeneic stem cell transplant with schedule that accommodates at least a 5 week exercise intervention, but not greater than 12 weeks
* Ability to understand and communicate in English
* Ability to understand and comply with study procedures for the entire length of the study
* Willing and able to provide written informed consent

Exclusion Criteria:

* Dementia, altered mental status, or psychiatric condition that would prohibit the understanding or rendering of informed consent
* Co-morbid illness that would contraindicate maximal effort exercise testing or participation in regular exercise programming as determined by the treating physician or exercise physiologist
* Concurrent radiation, chemotherapeutic, or investigational therapy other than transplant related therapy
* Concurrent enrollment in LCCC 1404

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Compare changes in VO2peak after a 5-12 week period of time prior to alloHCT in patients undergoing interval exercise training (IET) and motivational accelerometry (MA) vs patients receiving usual care (controls). | 5-12 weeks
  Patients will undergo a baseline fitness assessment consisting of cardiorespiratory exercise testing using indirect calorimetry on a cycle ergometer (for the assessment of VO2peak).

SECONDARY OUTCOMES:
Compare changes in 6 minute walk distance (6MWD) after a 5-12 week period of time prior to alloHCT in patients receiving IET/MA vs controls. | 5-12 weeks
Compare changes in peripheral blood p16INK4a after a 5-12 week period of time prior to alloHCT in patients receiving IET/MA vs controls. | 5-12 weeks

OTHER OUTCOMES:
Compare average steps per day during a 5-12 week period of time prior to alloHCT in patients receiving IET/MA vs. controls | 5-12 weeks
Compare post-alloHCT average steps per day in patients who received pre-alloHCT IET/MA vs controls. | Post-alloHCT refers to Day0 (transplant day) through Day+365
Compare post-alloHCT symptom burden and quality of life in patients who received pre-alloHCT IET/MA vs controls. | Post-alloHCT refers to Day0 (transplant day) through Day+365
Compare post-alloHCT days alive and out of the hospital within the first 100 days post-transplant in patients who received pre-alloHCT IET/MA vs controls. | Post-alloHCT refers to the initial discharge day after allo-HCT through the first 100 days out of the hospital and/or alive, whichever is the shorter duration.
Compare post-alloHCT survival in patients who received pre-alloHCT IET/MA vs controls. | Post-alloHCT refers to Day0 (transplant day) through Day+365

CONTACTS AND LOCATIONS:
Overall Officials: William A Wood, MD, MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bevans MF, Mitchell SA, Marden S. The symptom experience in the first 100 days following allogeneic hematopoietic stem cell transplantation (HSCT). Support Care Cancer. 2008 Nov;16(11):1243-54. doi: 10.1007/s00520-008-0420-6. Epub 2008 Mar 6. PMID 18322708
- [Background] Bevans M. Health-related quality of life following allogeneic hematopoietic stem cell transplantation. Hematology Am Soc Hematol Educ Program. 2010;2010:248-54. doi: 10.1182/asheducation-2010.1.248. PMID 21239801
- [Background] Khera N, Zeliadt SB, Lee SJ. Economics of hematopoietic cell transplantation. Blood. 2012 Aug 23;120(8):1545-51. doi: 10.1182/blood-2012-05-426783. Epub 2012 Jun 13. PMID 22700725
- [Background] Majhail NS, Rizzo JD, Hahn T, Lee SJ, McCarthy PL, Ammi M, Denzen E, Drexler R, Flesch S, James H, Omondi N, Pedersen TL, Murphy E, Pederson K. Pilot study of patient and caregiver out-of-pocket costs of allogeneic hematopoietic cell transplantation. Bone Marrow Transplant. 2013 Jun;48(6):865-71. doi: 10.1038/bmt.2012.248. Epub 2012 Dec 10. PMID 23222378
- [Background] Wiskemann J, Dreger P, Schwerdtfeger R, Bondong A, Huber G, Kleindienst N, Ulrich CM, Bohus M. Effects of a partly self-administered exercise program before, during, and after allogeneic stem cell transplantation. Blood. 2011 Mar 3;117(9):2604-13. doi: 10.1182/blood-2010-09-306308. Epub 2010 Dec 29. PMID 21190995
- [Background] Wiskemann J, Huber G. Physical exercise as adjuvant therapy for patients undergoing hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Feb;41(4):321-9. doi: 10.1038/sj.bmt.1705917. Epub 2007 Nov 19. PMID 18026154
- [Background] Nytroen K, Rustad LA, Aukrust P, Ueland T, Hallen J, Holm I, Rolid K, Lekva T, Fiane AE, Amlie JP, Aakhus S, Gullestad L. High-intensity interval training improves peak oxygen uptake and muscular exercise capacity in heart transplant recipients. Am J Transplant. 2012 Nov;12(11):3134-42. doi: 10.1111/j.1600-6143.2012.04221.x. Epub 2012 Aug 17. PMID 22900793
- [Background] Guiraud T, Labrunee M, Gaucher-Cazalis K, Despas F, Meyer P, Bosquet L, Gales C, Vaccaro A, Bousquet M, Galinier M, Senard JM, Pathak A. High-intensity interval exercise improves vagal tone and decreases arrhythmias in chronic heart failure. Med Sci Sports Exerc. 2013 Oct;45(10):1861-7. doi: 10.1249/MSS.0b013e3182967559. PMID 23591293
- [Background] Puhan MA, Busching G, Schunemann HJ, VanOort E, Zaugg C, Frey M. Interval versus continuous high-intensity exercise in chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2006 Dec 5;145(11):816-25. doi: 10.7326/0003-4819-145-11-200612050-00006. PMID 17146066
- [Background] Nybo L, Sundstrup E, Jakobsen MD, Mohr M, Hornstrup T, Simonsen L, Bulow J, Randers MB, Nielsen JJ, Aagaard P, Krustrup P. High-intensity training versus traditional exercise interventions for promoting health. Med Sci Sports Exerc. 2010 Oct;42(10):1951-8. doi: 10.1249/MSS.0b013e3181d99203. PMID 20195181
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Background] Shephard RJ. Tests of maximum oxygen intake. A critical review. Sports Med. 1984 Mar-Apr;1(2):99-124. doi: 10.2165/00007256-198401020-00002. PMID 6385195
- [Background] Jones LW, Eves ND, Haykowsky M, Joy AA, Douglas PS. Cardiorespiratory exercise testing in clinical oncology research: systematic review and practice recommendations. Lancet Oncol. 2008 Aug;9(8):757-65. doi: 10.1016/S1470-2045(08)70195-5. PMID 18672211
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Liu Y, Sanoff HK, Cho H, Burd CE, Torrice C, Ibrahim JG, Thomas NE, Sharpless NE. Expression of p16(INK4a) in peripheral blood T-cells is a biomarker of human aging. Aging Cell. 2009 Aug;8(4):439-48. doi: 10.1111/j.1474-9726.2009.00489.x. Epub 2009 May 22. PMID 19485966
- [Background] Sanoff HK, Deal AM, Krishnamurthy J, Torrice C, Dillon P, Sorrentino J, Ibrahim JG, Jolly TA, Williams G, Carey LA, Drobish A, Gordon BB, Alston S, Hurria A, Kleinhans K, Rudolph KL, Sharpless NE, Muss HB. Effect of cytotoxic chemotherapy on markers of molecular age in patients with breast cancer. J Natl Cancer Inst. 2014 Apr;106(4):dju057. doi: 10.1093/jnci/dju057. Epub 2014 Mar 28. PMID 24681605
- [Background] Hallal PC, Victora CG. Reliability and validity of the International Physical Activity Questionnaire (IPAQ). Med Sci Sports Exerc. 2004 Mar;36(3):556. doi: 10.1249/01.mss.0000117161.66394.07. No abstract available. PMID 15076800
- [Background] Wood WA, Deal AM, Bennett AV, Mitchell SA, Abernethy AP, Basch E, Bailey C, Reeve BB. Comparison of seven-day and repeated 24-hour recall of symptoms in the first 100 days after hematopoietic cell transplantation. J Pain Symptom Manage. 2015 Mar;49(3):513-20. doi: 10.1016/j.jpainsymman.2014.06.011. Epub 2014 Aug 13. PMID 25128608
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Angadi SS, Mookadam F, Lee CD, Tucker WJ, Haykowsky MJ, Gaesser GA. High-intensity interval training vs. moderate-intensity continuous exercise training in heart failure with preserved ejection fraction: a pilot study. J Appl Physiol (1985). 2015 Sep 15;119(6):753-8. doi: 10.1152/japplphysiol.00518.2014. Epub 2014 Sep 4. PMID 25190739
- [Background] Moholdt T, Bekken Vold M, Grimsmo J, Slordahl SA, Wisloff U. Home-based aerobic interval training improves peak oxygen uptake equal to residential cardiac rehabilitation: a randomized, controlled trial. PLoS One. 2012;7(7):e41199. doi: 10.1371/journal.pone.0041199. Epub 2012 Jul 18. PMID 22815970
- See also: Pasquini MC, Wang Z. Current use and outcome of hematopoietic stem cell transplantation: CIBMTR Summary Slides, 2011. Slides 3, 18, 21-40. — http://www.cibmtr.org
- See also: National Cancer Institute. Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). — http://healthcaredelivery.cancer.gov/pro-ctcae/
- See also: National Institutes of Health. Patient Reported Outcomes Measurement Information System (PROMIS). — http://www.nihpromis.org